CLINICAL TRIAL: NCT02446119
Title: Pyloric Sphincter Pressure and Geometry Assessment Using EndoFlip
Acronym: PyloEndoFlip
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 21560
Record Dates: First submitted 2015-05-09; First posted 2015-05-18 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastroparesis: Inclusion criteria:
  1. Subjects will be of either sex, 18 to 70 years of age.
  patients with an established diagnosis of gastroparesis, either diabetic or idiopathic etiology. The gastroparesis subjects will have delayed gastric emptying on gastric scintigraphy defined as greater than 60% retention at 2 hours and/or greater than 10% retention at 4 hours. This gastric emptying test would have been done prior to the endoscopy and is not part of the research study. Patients will undergo EndoFlip during upper endoscopy.
  Interventions: Device: EndoFLIP
- Normals: Inclusion criteria:
  1. Subjects will be of either sex, 18 to 70 years of age.
  control subjects will be nondiabetic patients without gastroparesis or gastroesophageal reflux symptoms undergoing upper endoscopy. Patients will undergo EndoFlip during upper endoscopy.
  Interventions: Device: EndoFLIP

INTERVENTIONS:
Device: EndoFLIP — Measurement of pyloric resistance and compliance

SUMMARY:
Gastroparesis is a disorder characterized by symptoms from gastric retention in the absence of mechanical obstruction. Gastric emptying is a highly regulated process reflecting the integration of the propulsive forces of proximal fundic tone and distal antral contractions with the functional resistance provided by the pyloric sphincter. Pylorospasm has been reported in some patients with gastroparesis. This study protocol will assess pyloric sphincter pressure and geometry in patients with gastroparesis and control subjects without symptoms of gastroparesis. The commercially available FDA approved endoscopic functional luminal imaging probe (EndoFLIP) catheter will be used, which measures diameter, pressure, length, and distensibility of gastrointestinal sphincter muscles along the balloon distance. It is used to measure the pressure characteristics of the lower esophageal sphincter during bariatric surgery for obesity, during Heller myotomy for achalasia, and during Nissen fundoplication for gastroesophageal reflux disease. In this study, during upper endoscopy, which is routinely performed under sedation, patients with gastroparesis and controls without gastroparesis symptoms will have their pyloric sphincter assessed with EndoFLIP. After passage of the endoscope into the stomach, the EndoFLIP catheter will be introduced alongside the endoscope and advanced through the pyloric sphincter as visualized endoscopically. The investigators will measure the pressure and contour of the pyloric sphincter using three successive volume distensions of the EndoFLIP balloon (20 ml, 30 ml, 40 ml). The investigators will compare the results between the gastroparesis patients and the control patients without gastroparesis. Through this study, the investigators will better understand the abnormalities of the pyloric sphincter in patients with gastroparesis.

DETAILED DESCRIPTION:
This study protocol will assess pyloric sphincter pressure and geometry in patients with gastroparesis and control subjects without symptoms of gastroparesis.

Aims: To determine if there is a subgroup of patients with gastroparesis who have pressure and/or geometric configuration abnormalities of the pyloric sphincter. We will determine this by assessing the pressure, diameter, length, and distensibility of the pyloric sphincter in patients with gastroparesis and in subjects without gastroparesis undergoing upper endoscopy for their clinical evaluation.

Hypothesis:The pylorus of patients with gastroparesis has a higher pressure, smaller diameter, and is less distensible than the pylorus of control patients without gastroparesis

Methods: The commercially available FDA approved endoscopic functional luminal imaging probe (EndoFLIP) catheter will be used, which measures diameter, pressure, length, and distensibility of gastrointestinal sphincter muscles along the balloon distance. It is used to measure the pressure characteristics of the lower esophageal sphincter during bariatric surgery for obesity, during Heller myotomy for achalasia, and during Nissen fundoplication for gastroesophageal reflux disease. In this study, during upper endoscopy, which is routinely performed under sedation, patients with gastroparesis and controls without gastroparesis symptoms will have their pyloric sphincter assessed with EndoFLIP. After passage of the endoscope into the stomach, the EndoFLIP catheter will be introduced alongside the endoscope and advanced through the pyloric sphincter as visualized endoscopically. The investigators will measure the pressure and contour of the pyloric sphincter using three successive volume distensions of the EndoFLIP balloon (20 ml, 30 ml, 40 ml). The assessment of the pylorus will be done during the upper endoscopy which will take approximately 60 minutes. We will compare the pyloric pressure measurements in patients with gastroparesis to the control patients. This is an observational study, with no intervention.

Analysis: The investigators will compare the results between the gastroparesis patients and the control patients without gastroparesis.

Through this study, the investigators will better understand the abnormalities of the pyloric sphincter in patients with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be of either sex, 18 to 70 years of age.
2. Two groups will be recruited:

   * First, patients with an established diagnosis of gastroparesis, either diabetic or idiopathic etiology.
   * Second, control subjects will be nondiabetic patients without gastroparesis or gastroesophageal reflux symptoms undergoing upper endoscopy.

Exclusion criteria Prior surgery involving the stomach

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  1. Subjects will be of either sex, 18 to 70 years of age.
  2. Two groups will be recruited. 2a. First, patients with an established diagnosis of gastroparesis, either diabetic or idiopathic etiology. The gastroparesis subjects will have delayed gastric emptying on gastric scintigraphy defined as greater than 60% retention at 2 hours and/or greater than 10% retention at 4 hours.
  2b. Second, control subjects will be nondiabetic patients without gastroparesis or gastroesophageal reflux symptoms undergoing upper endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-05; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pyloric pressure | 60 minutes
  Measurement of pyloric pressure using EndoFLIP in patients with gastroparesis and controls. Our plan is to compare the pyloric pressures in patients with gastroparesis to controls. This is an observational study with no intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Parkman, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States